CLINICAL TRIAL: NCT00234169
Title: A Phase I/II Study of Peripheral Blood Progenitor Cells Mobilisation With VTP195183 Plus G-CSF Compared to Mobilisation With G-CSF Alone in Patients With Multiple Myeloma and Lymphoma.
Brief Title: A Study of Peripheral Blood Progenitor Cells Mobilisation (PBPC) With VTP195183 Plus Granulocyte-Colony Stimulating Factor (G-CSF) Compared to Mobilisation With G-CSF Alone
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, Kirsten Herbert, Doctor, Peter MacCallum Cancer Centre, Australia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/09
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Multiple Myeloma; Lymphoma
Keywords: Multiple Myeloma; Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: VTP195183 — VTP195183: 60mg/m2 orally daily G-CSF: 10mcg/kg/day subcutaneously Provision is made for dose reduction of VTP195183 in the event of unexpected dose-limiting toxicities G-CSF10mcg/kg/day will commence on day 1 and will continue until the peripheral blood (PB) CD34+ count falls below baseline, or below 5 x 106/L, whichever happens first.
  Patients will be treated with VTP195183 alone at 60mg/m2/day from day 1 to day 7. On day 8 VTP195183 will be continued and G-CSF10mcg/kg/day will be added. VTP195183 plus G-CSF will continue until the peripheral blood (PB) CD34+ count falls below baseline, or below 5 x 106/L, whichever happens first.

SUMMARY:
Hematopoietic stem cells (HSC) are used to support the administration of high dose chemotherapy for a range of human cancers. For a safe HSC transplantation, a minimum of 5 million HSC per kilogram are required. HSC are collected from the bone marrow by using drugs such as G-CSF (filgrastim) which 'mobilize' them from the bone marrow into the bloodstream. HSC are collected from the bloodstream using an apheresis machine. Between 5 and 60% of patients fail to mobilize the minimum HSC dose required for safe transplantation, and this trial is investigating a way to enhance mobilization to overcome this problem. This trial aims to determine if a new vitamin A derivative is capable of enhancing HSC mobilization when used in conjunction with G-CSF. Patients will undergo two mobilization procedures. They will be given G-CSF alone, or a combination of the study drug plus G-CSF, and their stem cells will be collected. A comparison group of patients will be given G-CSF alone for both mobilizations. Stem cells collected from patients in this trial will be frozen and stored until they are required for transplantation into that patient. At that time, patients will be monitored for how well they recover from their high dose chemotherapy and HSC transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70
2. Histologically proven multiple myeloma or lymphoma
3. Intent of treating physician to proceed to high dose therapy and autologous transplantation
4. Not currently receiving thalidomide (within 1 week of commencing VTP195813 or G-CSF), cytotoxic agents or high dose prednisolone or Dexamethasone (at doses greater than 15 mg prednisolone or equivalent per day)
5. Multiple myeloma patients must be taking regular bisphosphonate therapy
6. Absolute neutrophil count between 1.5 and 10 x 109/L
7. ECOG performance status ? 2
8. Life expectancy of at least 2 months
9. Written informed consent signed by patient or legally authorized representative

Exclusion Criteria:

1. Active infection or a fever > 38.2 degrees C (fever due to B symptoms in lymphoma patients will not exclude a patient)
2. Use within the previous 30 days of other vitamin A preparations within the last 30 days (including oral vitamin supplements, oral retinoids for acne or other skin disorders, bexarotene, or topical vitamin A preparations)
3. Pregnancy or breast feeding. Women of child-bearing potential, admitted to the trial must take adequate measures to prevent conception (at least two different forms of contraception during the study and for at least one month after completion of study drugs) and are to undergo a pregnancy test
4. Significant non-malignant disease including HIV infection, uncontrolled hypertension (diastolic blood pressures > 115 mmHg), unstable angina
5. Known allergy to E.coli-derived products
6. Current treatment with tetracycline antibiotics

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
PB CD34+ kinetics using VTP195183 plus G-CSF | up to 28 days post study drug administration

SECONDARY OUTCOMES:
The toxicity of VTP195183 pretreatment when used with G-CSF | within 28 days of study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Herbert, MBBS, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer centre, Melbourne, Victoria, Australia